CLINICAL TRIAL: NCT06474910
Title: Connective Tissue Massage in Patients With Scleroderma
Brief Title: Connective Tissue Massage in Scleroderma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Head of Physiotherapy and Rehabilitation Department, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/07-34
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Scleroderma
Keywords: Scleroderma; Connective tissue massage; mobility
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective tissue massage group (Experimental): In addition to the exercise program for hand rehabilitation, 15 patients in this group will receive connective tissue massage of the hand and forearm area. The exercise program will include stretching exercises for the hand, strengthening exercises, normal joint movement exercises, functional exercises and tendon sliding exercises.
  Interventions: Other: Connective tissue massage
- Exercise group (Experimental): Only exercise program will be applied to 15 patients in this group. The exercise program will include stretching exercises for the hand, strengthening exercises, normal joint movement exercises, functional exercises and tendon sliding exercises.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Connective tissue massage — In addition to the exercise program for hand rehabilitation, 15 patients in this group will receive connective tissue massage of the hand and forearm area. The exercise program will include stretching exercises for the hand, strengthening exercises, normal joint movement exercises, functional exercises and tendon sliding exercises.
  Arms: Connective tissue massage group
Other: Exercise — Only exercise program will be applied to 15 patients in this group. The exercise program will include stretching exercises for the hand, strengthening exercises, normal joint movement exercises, functional exercises and tendon sliding exercises.
  Arms: Exercise group

SUMMARY:
The only study in the literature that examined connective tissue massage in patients with scleroderma is by Bongi et al. In this study, connective tissue massage and Mc Mennell joint manipulation technique were applied to the experimental group in addition to the home exercise program. The control group was offered only a home exercise program. The results of the study showed that the group in which connective tissue massage and Mc Mennell joint manipulation technique were applied were effective on hand functions, quality of life and mobility. The aim of our study was to examine the effects of connective tissue massage applied in addition to the exercise program.The study will include 30 patients diagnosed with scleroderma according to American College of Rheumatology/European League Against Rheumatism criteria and followed up in Fırat University Rheumatology Department. Patients will be divided into two groups; 15 patients in the first group will be applied connective tissue massage to the hand and forearm area in addition to the exercise program for hand rehabilitation. In the second group, 15 patients will only receive an exercise program.

DETAILED DESCRIPTION:
Although there are various physiotherapy interventions in scleroderma rehabilitation, there is no definitive guideline. Passive and active stretching has been shown to help maintain range of motion (ROM) and optimal length of structures. Home exercises form part of rehabilitation in most studies. The only study in the literature that examined connective tissue massage in patients with scleroderma is by Bongi et al. In this study, connective tissue massage and Mc Mennell joint manipulation technique were applied to the experimental group in addition to the home exercise program. The control group was offered only a home exercise program. The results of the study showed that the group in which connective tissue massage and Mc Mennell joint manipulation technique were applied were effective on hand functions, quality of life and mobility. The aim of our study was to examine the effects of connective tissue massage applied in addition to the exercise program.The study will include 30 patients diagnosed with scleroderma according to American College of Rheumatology/European League Against Rheumatism criteria and followed up in Fırat University Rheumatology Department. Patients will be divided into two groups; 15 patients in the first group will be applied connective tissue massage to the hand and forearm area in addition to the exercise program for hand rehabilitation. In the second group, 15 patients will only receive an exercise program. Range of motion, skin thickness and hand mobility test will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Stable on medical treatment
* Be able to adapt to exercise

Exclusion Criteria:

* Diagnosed with juvenile onset scleroderma
* Accompanied by another rheumatic disease
* Active digital ulcer
* Chronic disease or trauma history that will affect hand functions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-21 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Mobility assessment | 2 minutes
  The hand function test developed for SSc patients will be used to assess specific functions of the patients. The ability to use the hand in daily tasks and limitation of movement will be evaluated. Finger movements, grasping, releasing, pronation, supination movements are scored between 0-3.

SECONDARY OUTCOMES:
Skin thickness assessment | 1 minute
  The modified Rodnan skin score (mRSS) will be used to assess skin thickness. Normal skin thickness will be scored as zero, mild skin thickening as one, difficulty in making skin folds and wrinkle-free skin thickness as two, inability to hold the skin between two fingers and severe skin thickness as three.
Range of motion assessment | 2 minutes
  The ROM of the fingers will be measured with a finger goniometer. Distal interphalangeal (DIP), proximal interphalangeal (PIP) and metacarpophalangeal (MCP) joint flexion ranges of motion will be measured with the forearm and wrist in neutral position and fingers in maximum flexion (fist position).

CONTACTS AND LOCATIONS:
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No